CLINICAL TRIAL: NCT01174589
Title: Strength Training of Patients With Hip Fracture - a Randomized Clinical Trial
Brief Title: Training of Patients With Hip Fracture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lolland Community, Denmark (Other)
Collaborators: Association of Danish Physiotherapists (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mr. Jan Overgaard, Physiotherapist, Bachelor, Sector of Health, Rehabilitation, Lolland Community., Lolland Community, Denmark
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-145
Record Dates: First submitted 2010-07-21; First posted 2010-08-03 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hip Fracture
Keywords: Lower limb strength training; Randomized clinical trial; Patients with Hip fracture; 6 vs. 12 weeks physical strength training
MeSH Terms: conditions — Hip Fractures | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 weeks of physical training (Other): The 6 weeks of physical training consists of muscle strength training of both legs, balance and coordination exercises 2 times a week.
  Interventions: Other: Strength training
- 12 weeks of physical exercise (Other): The 12 weeks of physical training consists of muscle strength training of both legs, balance and coordination exercises 2 times a week.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — to compare if there is a difference between 6 or 12 weeks of physical strength training

SUMMARY:
The primary purpose of this study is to illustrate whether there is a difference in the 6 minutes walking test in patients with hip fractures who have received 6 vs. 12 weeks of physical training after discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip fractures
* full weightbearing on the affected leg
* patients living in their own home with an independent walking ability score >=2 according to the New Mobility Score scale
* written consent

Exclusion Criteria:

* institutionalized patients
* more than 2 weeks after discharge from hospital
* non weight bearing on the affected leg
* Dementia
* other conditions/diagnosis that would have an effect on the ability to train eg. neurological diagnosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference in the 6-minutes walking test | at baseline, 6 weeks, 12 weeks (primary analysis) and 24 weeks after baseline testing
  The 6-minutes walking test, performed according to international guidelines.

SECONDARY OUTCOMES:
Difference of the Maximal isometric knee-extension strength of the fractured limb. | Baseline, 6 weeks, 12 weeks and 24 weeks after baseline testing
  The best of 5 maximal isometric unilateral knee-extension strength tests of both limbs, measured with a fixated handheld dynamometer
Difference in 10-meter fast speed walking test | At baseline, 6 weeks, 12 weeks, and 24 weeks after baseline testing
  Best of 3 timed 10 meter fast speed walk tests.
Difference in the Timed Up & Go test | At baseline and 6 weeks, 12 weeks and 24 weeks after baseline testing
  Best of 3 timed TUG tests will be used.
Difference in the Short Form-36 | At baseline, 6 weeks, 12 weeks and 24 weeks after baseline testing
  The Questionnaire will be filled out during an interview with the patient
Difference in the New Mobility Score | At baseline, 6 weeks, 12 weeks and 24 weeks after baseline testing
  The questionnaire will be filled out during an interview with the patient.

OTHER OUTCOMES:
Difference in the Barthel 0-20 points ADL-score | At baseline, 6 weeks, 12 weeks and 24 weeks after baseline testing
  The questionnaire will be filled out during an interview with the patient
The Tandem Balance test 0-30 points | At baseline, 6 weeks, 12 weeks and 24 weeks after baseline testing

CONTACTS AND LOCATIONS:
Overall Officials: Jan Overgaard, MSc., Principal Investigator — Sector of health, rehabilitation, Lolland community, Denmark; Morten T Kristensen, PhD, Study Director — Department of Physical Therapy and Orthopedic Surgery, Copenhagen University Hospital at Hvidovre, Denmark
Locations (1):
- Maribo Health Center, Maribo, Denmark

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Overgaard JA, Kallemose T, Mangione KK, Kristensen MT. Six Versus 12 Weeks of Outpatient Physical Therapy Including Progressive Resistance Training in Cognitively Intact Older Adults After Hip Fracture: A Multicenter Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2022 Jul 5;77(7):1455-1462. doi: 10.1093/gerona/glab256. PMID 34460897